CLINICAL TRIAL: NCT00569868
Title: UARK 2005-05, Coagulation-Related Effects of Velcade Treatment in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Bart Barlogie, MD, PhD, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2005-05
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-07

CONDITIONS: MULTIPLE MYELOMA
Keywords: PLASMACYTOMA
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade (Experimental): Treatment on this study will last 2 cycles. Each cycle consists of 3 weeks, or 21 days. After you have gone off study, you will be followed every three months for approximately 2 years.
  Each cycle will consist of 3 weeks (21 days) according to the schedule below.
  DRUG ROUTE DOSE DAYS Velcade IV 1.3 mg/m2 1,4,8, and 11 This 21-day period will be considered one treatment cycle; Cycle 2 would commence on Day 22 (Cycle 2, Day 1). Patients may continue to receive treatment every 21 days, provided there is no evidence of disease progression or no unacceptable toxicity for a two cycles.
  Interventions: Drug: Velcade

INTERVENTIONS:
Drug: Velcade — Except for the two PCR-based genotyping assays, which will be conducted only on baseline samples, tests will be assessed at baseline, 1-3 hours after the first dose of Velcade day 1 and on day 11 of the first cycle of Velcade.
  The platelet Aggregation Test will be done only if Platelet count is 100 000.

SUMMARY:
To evaluate changes in coagulation (blood clotting) factors and platelet function in multiple myeloma participants undergoing VELCADE treatment for the first time.

DETAILED DESCRIPTION:
Cardiovascular complications during the treatment of patients with multiple myeloma are not uncommon, (10%) and the frequency clearly increases with the use of regimens containing thalidomide in combination with glucocorticosteroids or chemotherapy especially adriamycin. Even with prophylactic anticoagulation, DVT still occurs in 10% of such patients. The use of full anticoagulation raises considerable concern of bleeding especially during the post chemotherapy thrombocytopenic period. We observed no thromboembolic episodes when Velcade was added to thalidomide and adriamycin containing chemotherapy.

Therefore, we would like to investigate this protective antithrombotic effect of VELCADE in a malignancy associated with a hypercoagulable state in a group of 10 patients with Relapsed/Refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myeloma who had relapsed after one prior treatment and who have demonstrated resistance to their last treatment, who are candidate to receive Velcade and had normal PT and PTT, will be evaluated for inclusion in the present study.

Exclusion Criteria:

* Previous history of venous thromboembolism, myocardial infarction, stroke, TIA
* Hypercoagulable state (deficit ATIII, Factor V Leiden, deficit protein S, deficit protein C, prothrombin gene mutation), antiphospholipid syndrome.
* Von Willebrand disease, inherited platelet abnormalities.
* Familiar history of hypercoagulable state.
* Anticoagulant therapy, aspirin, non-steroidal anti-inflammatory drugs, beta blockers, tricyclic antidepressant, hormone replacement therapy, BCPs, and all other agents able to interfere with platelet function in the previous two weeks.
* Non-secretory MM, unless the patient has measurable lesions on CT, MRI and/or PET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Zangari M, Yaccoby S, Pappas L, Cavallo F, Kumar NS, Ranganathan S, Suva LJ, Gruenwald JM, Kern S, Zhan F, Esseltine D, Tricot G. A prospective evaluation of the biochemical, metabolic, hormonal and structural bone changes associated with bortezomib response in multiple myeloma patients. Haematologica. 2011 Feb;96(2):333-6. doi: 10.3324/haematol.2010.031302. Epub 2010 Oct 15. PMID 20952514
- See also: Myeloma Institute for Research and Therapy — http://www.myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade: Velcade IV, 1.3 mg/m2, days 1,4,8, and 11: Treatment on this study will last 2 cycles. Each cycle consists of 3 weeks, or 21 days, then followed every three months for approximately 2 years.
Period: Overall Study
Arm/Group | Velcade
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Velcade
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Antithrombotic Effect of VELCADE in a Malignancy Associated With a Hypercoagulable State in Patients With Relapsed/Refractory Multiple Myeloma.
Description: Goal is to evaluate changes in coagulation (blood clotting) in refractory/relapsing multiple myeloma patients during VELCADE treatment.
  Before and during treatment, participant will undergo routine tests/procedures following the Myeloma Institute's guidelines (physical exams, blood, urine, and bone tests, and bone marrow aspirates and biopsies) and will also receive a series of coagulation tests before treatment and after 1st and 3rd doses of each cycle.
  Response measured as: complete, partial, or minimal response, no change, progressive disease, or relapse from complete response.
Time Frame: 60 days
Population: no analysis done, descriptive information on the magnitude, direction, and variability of changes in coagulation factors and platelet function in refractory/relapsing multiple myeloma patients during VELCADE treatment was collected
Measure: Number; unit: participants
Arm/Group | Velcade
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Velcade
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No